CLINICAL TRIAL: NCT05790941
Title: Proof of Concept of Latanoprost/Minoxidil (ANR-001.1) Topical Formulation for Eyebrows
Brief Title: Proof of Concept Study of Latanoprost/Minoxidil (ANR-001.1) Topical Formulation
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aneira Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ANR C001
Record Dates: First submitted 2023-03-17; First posted 2023-03-30 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-02

CONDITIONS: Hypotrichosis
Keywords: Eyebrow
MeSH Terms: conditions — Hypotrichosis | interventions — Latanoprost; Minoxidil

STUDY DESIGN:
Who Masked: Participant
Masking Description: Unlabeled bottle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Latanoprost/Minoxidil formulation (Experimental): 8 participants: Topical Latanoprost/Minoxidil formulation applied to both eyebrows once a day for 90 days
  Interventions: Combination Product: Latanoprost and Minoxidil
- Control Group (Placebo Comparator): 4 participants: Vehicle applied to both eyebrows once a day for 90 days
  Interventions: Combination Product: Latanoprost and Minoxidil

INTERVENTIONS:
Combination Product: Latanoprost and Minoxidil — Latanoprost and Minoxidil formulation for the treatment of hypotrichosis of the eyebrows.

SUMMARY:
Study to Evaluate the safety and efficacy of a Latanoprost/Minoxidil formulation vs. placebo for the treatment of hypotrichosis of the eyebrows.

DETAILED DESCRIPTION:
A Single-Blind placebo controlled trial of the efficacy and safety of the treatment of hypotrichosis of the eyebrows comparing a subset of patients receiving a combination of latanoprost/minoxidil formulation as compared to placebo measured by a validated imaging system.

ELIGIBILITY:
Inclusion Criteria: • Subjects, age 22 to 65 years, in general good health.

* Patients with diagnosed hypotrichosis of the eyebrows.
* Subjects with active hair loss within the last 12 months.
* Patients willing to refrain from initiation of any new vitamins or nutritional supplements for the duration of the study.
* Patients willing to refrain from use of any hair growth therapies (oral or topical) other than the investigational product.

Exclusion Criteria: • Subjects with an active disease or infection, or chronic dermatological condition (eczema, psoriasis, infection, etc.) of the scalp that may interfere with the assessment of scalp skin health in the treated regions.

* History of hair transplants, scalp reduction, current hair weave or tattooing in the target area, artificial hair coloring two months prior to initiation of study which makes it difficult to perform hair count assessment.
* Subjects with hair loss for greater than 5 years, as medical therapy is unlikely to have much effect at restoring hair follicles inactive for that long of a time period.
* Subjects with a history of chemotherapy, receiving cytotoxic agents, radiation, or laser/surgical therapy of the scalp within the past 12 months.
* Any known or underlying medical problem that could influence hair growth such as HIV infection, connective tissue disease, a thyroid condition, inflammatory bowel disease or other medical conditions, at the discretion of the investigator.
* Subjects with clinical diagnosis of hair loss other than hypotrichosis of the eyebrows.
* Subjects with severe cardiovascular disease, uncontrolled or untreated hypertension, arrythmia or clinically relevant hypotension.
* Subjects with known or suspected hypersensitivity or allergic reaction to any of the active or inactive components of the test articles.
* Pregnant or lactating females or planning to become pregnant for the duration of the study.
* Subjects using medications that potentially cause drug-induced hair loss (e.g., depotestosterone, haloperidol, methotrexate, methylprednisolone, prednisone, testosterone, divalproex sodium) within the last 3 months.
* Current enrollment in any other investigational medication (drug) study within the 4 weeks prior to study initiation.
* Current or recent (2 months) history of severe diet or eating disorder.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-03-11 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Target Area Hair Count | 90 days
  Target Area Hair Count as Determined by the Brigham Tool for Alopecia

SECONDARY OUTCOMES:
Standardized Global Photographs | 90 days
  1. Standardized Global Photographs and change from baseline measurement of eyebrow hair fullness using Canfield Eyebrow Hair Image Analysis.
Change in Total Area Hair Darkness | 90 days
  2. Change in Total Area Hair Darkness of non-vellus hairs as compared to baseline in target area, defined as change from baseline of non-vellus hairs measured in intensity units as determined by Canfield Eyebrow Hair Image Analysis.

OTHER OUTCOMES:
Subject Self Assessment | 90 Days
  1. Subject Self-Assessment and Investigator Global Assessment using a Canfield side-by-side comparison tool on Day 90. Measure participant's satisfaction with eyebrow treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dan Cosgrove, M.D., Principal Investigator — WellMax
Locations (1):
- WellMax, Indian Wells, California, United States

IPD SHARING:
Plan to Share IPD: No